CLINICAL TRIAL: NCT01010984
Title: Transcatheter Arterial Chemoembolization With Doxorubicin-loaded LC Beads in the Treatment of Liver-dominant Metastases in Patients With Stage IV Metastatic Melanoma
Brief Title: LC Bead Embolization Agent With Doxorubicin in the Treatment Liver Metastasis From Melanoma
Acronym: DEBDOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert C. Martin (Other)
Collaborators: University of Louisville (Other); Thomas Jefferson University (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Robert C. Martin, Professor University of Louisville, University of Louisville
Organization: University of Louisville (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G090097
Record Dates: First submitted 2009-11-04; First posted 2009-11-10 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-03

CONDITIONS: Stage IV Melanoma
Keywords: metastatic melanoma; stage IV melanoma; metastatic melanoma to the liver
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcatheter Arterial Chemoembolization (Experimental): TACE using LC beads loaded with Doxorubicin
  Interventions: Device: LC beads loaded with Doxorubicin

INTERVENTIONS:
Device: LC beads loaded with Doxorubicin — During each TACE, 2 vials (1 vial, 75mg Doxorubicin) of 100-300 micrometer size LC beads loaded with doxorubicin will be delivered to the liver tumor(s). Total Doxorubicin dose for each TACE is 150mg

SUMMARY:
The purpose of this study is to determine if LC beads loaded with Doxorubicin are a safe and effective treatment for melanoma that has spread to the liver.

DETAILED DESCRIPTION:
In this study, trans-arterial chemoembolization will be used to deliver LC beads loaded with Doxorubicin directly into liver tumors resulting from malignant melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable, measurable disease defined as at least one lesion that can be accurately and serially measured per the modified RECIST and EASL criteria (2D/3D-EASL) or MRI (Extent of Necrosis)
* Patients ≥ 18 years of age, > 35kg, of any race or sex, who have histological or radiological proof of melanoma to the liver
* ECOG performance status < 3
* Patient chooses to participate and has signed the informed consent document
* Patients with unilobar disease who can be treated superselectively in a single session or patients with bilobar disease who can have both lobes able to be treated within 3 - 4 weeks in separate sessions
* Patients with patent main portal vein
* Ocular melanoma is allowed
* Patients with clinically and radiologically stable brain metastasis from melanoma can be included
* Patients with liver dominant disease (>50% overall tumor burden)
* Prior systemic therapy for metastatic disease is allowed
* Non-pregnant with an acceptable contraception in premenopausal women and fertile men
* Hematological function: ANC ≥1.5 x 109/L, platelets ≥ 75 x 109/L, INR ≤1.3 (patients on therapeutic anticoagulants are not eligible)
* Adequate renal function: Creatinine ≤2.0mg/dl and GFR >30
* Adequate liver function: total bilirubin ≤ 2.5 mg/dl, ALT, AST ≤ 5 times ULN, albumin ≥ 2.5mg/dl
* All toxic effects of prior therapy must have resolved to ≤ Grade 1 unless otherwise specified above

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Patients eligible for curative treatment such as resection or radiofrequency ablation
* Active bacterial, viral or fungal infection within 72 hours of study entry
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (TA, Tis & Ti) or any cancer curatively treated < 5 years prior to study entry
* Contraindication to hepatic artery embolization procedures:
* Severe peripheral vascular disease precluding catheterization
* Large shunt as determined by the investigator (pretesting with TcMAA not required) at the time of first angiogram
* Hepatofugal blood flow
* Main portal vein occlusion (e.g. thrombus or tumor)
* Recovery from major trauma including surgery within 4 weeks prior to administration of study treatment.
* Allergy to contrast media that cannot be managed with standard care (e.g. steroids), making magnetic resonance imaging (MRI) or computed tomography (CT) contraindicated
* Advanced liver disease (> 80% liver replacement)
* Other significant medical or surgical condition, or any medication or treatment that would place the patient at undue risk and that would preclude the safe use of chemoembolization or would interfere with study participation
* Any contraindication for doxorubicin administration:
* WBC <3000 cells/mm3
* Neutrophils <1500 cells/mm3
* Deficient cardiac function defined as a LVEF of <50% normal

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert CG Martin, MD, PhD, Study Director — University of Louisville
Locations (3):
- United States (3):
  - University of Louisville, Louisville, Kentucky
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Rostas JW, Tam AL, Sato T, Scoggins CR, McMasters KM, Martin RCG 2nd. Health-related quality of life during trans-arterial chemoembolization with drug-eluting beads loaded with doxorubicin (DEBDOX) for unresectable hepatic metastases from ocular melanoma. Am J Surg. 2017 Nov;214(5):884-890. doi: 10.1016/j.amjsurg.2017.07.007. Epub 2017 Jul 21. PMID 28754534
- [Derived] Rostas J, Tam A, Sato T, Kelly L, Tatum C, Scoggins C, McMasters K, Martin RCG 2nd. Image-Guided Transarterial Chemoembolization With Drug-Eluting Beads Loaded with Doxorubicin (DEBDOX) for Unresectable Hepatic Metastases from Melanoma: Technique and Outcomes. Cardiovasc Intervent Radiol. 2017 Sep;40(9):1392-1400. doi: 10.1007/s00270-017-1651-z. Epub 2017 May 15. PMID 28508253

RESULTS

PARTICIPANT FLOW:
Groups:
- Tace Using LC Beads Loaded With 150mg of Doxorubicin: Tace using LC beads loaded with 150mg of Doxorubicin. May have up to 6 treatments.
Period: Overall Study
Arm/Group | Tace Using LC Beads Loaded With 150mg of Doxorubicin
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transcatheter Arterial Chemoembolization
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Adverse events were collected from all 20 subjects.
Time Frame: Date of surgery through 2 years post procedure or until patient death
Population: Participants who received at least one dose of LC beads with doxorubin.
Measure: Number; unit: Events
Groups:
- Single Arm: Tace using LC beads loaded with 150mg of Doxorubicin. May have up to 6 treatments.
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Events | 465

2. Secondary Outcome: Percentage of Tumor Response
Description: Progression is determined using Modified Response Evaluation Criteria in Solid Tumors (mRECIST). Progressive disease is defined as at least 20% increase in the sum of the longest target lesions, taking as reference the smallest sum longest diameter recorded since start of treatment OR appearance of one or more new lesions greater then 1cm in size. Percentage of tumor response will be assessed up to 1 year post treatment.
Time Frame: Percentage of tumor response assessed up to 1 year post treatment.
Population: Those who receive at least one dose of LC bead with doxorubin.
Measure: Median (95% Confidence Interval); unit: percentage of tumor response
Groups:
- Tace Using LC Beads Loaded With Doxorubicin: Tace using LC beads loaded with 150mg doxorubicin. Treatment repeats every 3-4 weeks. Two to three treatments may be had in each lobe of the liver.
Arm/Group | Tace Using LC Beads Loaded With Doxorubicin
Number analyzed (Participants) | 20
percentage of tumor response | 2.46 [1.48 to 3.48]

ADVERSE EVENTS:
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 19/20
Serious Adverse Events (participants affected / at risk) | 19/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=20)
Hepatic Biliary Dilitation (Hepatobiliary disorders) | 3 (3)
Intractable Nausea (Gastrointestinal disorders) | 3 (3)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Enteritis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Ruptured Hepatic Lesion (Hepatobiliary disorders) | 1 (1)
Perforated Bowel (General disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Staph Infection (Infections and infestations) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Over Sedation (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=20)
Constipation (Gastrointestinal disorders) | 14 (14)
Peripheral Edema (General disorders) | 3 (3)
Weight Gain (Investigations) | 1 (1)
Weight Loss (Investigations) | 3 (3)
Hyperbilirubinemia (Investigations) | 1 (1)
Hypertension (Investigations) | 1 (1)
Penile Swelling (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal Burning Sensation (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Lack of Appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional State (Psychiatric disorders) | 2 (2)
Hallucinations (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Somnolence (Psychiatric disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Sinus Congestion (Immune system disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Bile Duct Necrosis (Hepatobiliary disorders) | 2 (2)
Ocular Icterus (Hepatobiliary disorders) | 1 (1)
Biliary Dilitation with Biloma (Hepatobiliary disorders) | 1 (1)
Biliary Dilatation (Hepatobiliary disorders) | 1 (1)
Biloma (Hepatobiliary disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Musculoskeletal Pain Chest (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood Pressure Increased (Investigations) | 2 (2)
Blood Bilirubin Increased (Investigations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Fungal Skin Infection (Infections and infestations) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
Thrombophlebitis (Vascular disorders) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (4)
Lethargy (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Tremor (Nervous system disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No